CLINICAL TRIAL: NCT05082467
Title: Prolonged Cardiac Patch Ambulatory Electrocardiogram Versus Conventional Holter Recording For Detection of Atrial Fibrillation After Cerebral Ischemic Event: A Comparative Analysis
Brief Title: Prolonged Cardiac ECG Patch Versus Conventional Holter For Detecting Atrial Fibrillation After Cerebral Ischemic Event
Acronym: PROVE-AF
Status: Active, not recruiting | Type: Observational
Sponsor: Sarawak General Hospital (Other)
Collaborators: Sarawak Heart Centre (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Diana Hui Ping Foo, Principal Investigator, Sarawak General Hospital
Other Study IDs: NMRR-19-3798-52441
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Stroke; Atrial Fibrillation; Cardiac ECG Patch
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to compare the diagnostic yield of water-resistant, wireless 7-day cardiac ECG patch versus conventional 24-hour Holter recording in detecting paroxysmal atrial fibrillation in patients admitted with acute ischemic stroke or transient ischemic attack of undetermined etiology after completion of a standard clinical stroke workup.

DETAILED DESCRIPTION:
This is a cohort study with a paired comparison between a cardiac ECG patch and conventional Holter system to detect atrial fibrillation in patients with acute ischemic stroke or transient ischemic attack of undetermined etiology. An estimated total of 320 adult patients will be enrolled in this study. Each eligible patient will receive simultaneously a conventional 24h Holter monitoring and a 7d cardiac ECG patch monitoring.

OBJECTIVES:

Primary objective:

To determine the diagnostic yield of a cardiac ECG patch compared to conventional Holter monitor for detecting occult paroxysmal atrial fibrillation (AF) within 24 hours in patients admitted with acute ischemic stroke or transient ischemic attack (TIA) of undetermined etiology after completion of a standard clinical stroke work-up.

Secondary objective(s):

* To determine efficacy of prolonged 7-day ambulatory ECG monitoring (using cardiac ECG patch) compared to conventional 24-hour ambulatory ECG monitoring (using conventional Holter) strategies in detecting paroxysmal AF.
* To determine if a strategy of a prolonged 7-day ambulatory ECG monitoring results in a change in clinical practice, i.e., more patients are anticoagulated.
* To assess the time to the first detection of AF within the first 7 days of monitoring.

Exploratory objective(s):

* To identify predictors of occult AF based on clinical, neuroimaging, echocardiography, and ECG features.
* To assess feasibility and cost-effectiveness of 7-day cardiac ECG patch monitoring for detecting occult paroxysmal AF.

SCREENING:

* Written informed consent obtained from patient or guardian
* Inclusion/Exclusion criteria.
* Social demographics, Risk factors, Comorbidities, Admission Brain CT/MRI,Stroke status including date and time of index event, date and time of admission, admission modified Rankin scale/NIHSS Score [Data extracted from patient records].
* 12-lead ECG, Transthoracic Echocardiogram

Eligible patients will be enrolled in the study and proceed with a baseline assessment.

BASELINE ASSESSMENT:

* Concomitant medication, Oxfordshire classification of stroke and CHA2DS2VAS Score [Data extracted from patient records].
* Anthropometric measurements and vital signs assessments
* 24h Holter and 7d Cardiac ECG patch monitoring

FOLLOW UP VISITS:

Follow-up visits will occur at 3 months and 1 year for the efficacy and outcomes for the duration of the study. There will be a total of 2 visits.The investigator/study team will perform the following procedures at each visit where applicable:

* Clinical examination (NIHSS Score assessment)
* Review concomitant medications
* AE/SAE assessment and monitoring
* Outcomes assessment
* Health outcome interview with EQ-5D Questionnaire
* TOAST Classification (at 1 year follow up visit)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Diagnosis of acute ischemic stroke or transient ischemic attack (TIA) (WHO definition) of undetermined etiology made by neurologist within 7 days after the index event. The event must be either:

   * an ischemic stroke confirmed by neuroimaging; or
   * a TIA, defined as involving a focal unilateral motor deficit, speech/language deficit or hemianopia, with symptom duration <24 hours (note: amaurosis fugax/ transient monocular blindness, pure sensory spells, isolated vertigo spells, etc. do not qualify for enrolment given the potential for misdiagnosis of such events).
3. No AF detected in baseline 12-lead ECG on admission.
4. The following diagnostic test have already been completed as part of clinical routine post-stroke/TIA:

   * Brain imaging with CT or MRI,
   * Transthoracic echocardiography to congenital heart disease and endocarditis.
5. Recurrent stroke/TIA is inclusionary as long as patient meets inclusion/exclusion criteria for study enrolment.

Exclusion Criteria:

1. Stroke of unknown time of symptom onset.
2. Modified Rankin Scale ≥5 on index admission.
3. Previous documented history of primary intracerebral bleeding.
4. Previous documented history of AF or atrial flutter (a remote history of transient AF during perioperative period is not exclusionary).
5. Skin allergies, conditions, or sensitivities to cardiac patch.
6. Exclusively retinal stroke or retinal TIA event.
7. Pre-existing indication for anticoagulation (eg. History of mechanical heart valve replacement, deep vein thrombosis).
8. Pre-existing contraindication for permanent anticoagulation (eg. hypocoagulable state).
9. Echocardiographic findings of congenital heart disease and endocarditis.
10. Indicated for pacemaker, implantable cardiac defibrillator (ICD), CRT device, or an implantable hemodynamic monitoring system.
11. Intravenous drug users (IVDUs).
12. Life expectancy < 1 year for reasons other than stroke (eg. Metastatic cancer disease).
13. Concomitant participation in other clinical trials involving investigational medications.
14. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are admitted with acute ischemic stroke or transient ischemic attack (TIA) of undetermined etiology after completion of a standard clinical stroke work-up will be included.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of newly diagnosed AF or atrial flutter within 24 hours of monitoring with cardiac ECG patch compared to conventional Holter. | 24 hours
  Detection of newly diagnosed AF or atrial flutter within 24 hours of monitoring with cardiac ECG patch compared to conventional Holter.

SECONDARY OUTCOMES:
Detection of AF or atrial flutter within 7 days of monitoring. | 7 days
  Detection of one or more episodes of AF or atrial flutter as assessed after 7 days of Holter monitoring.
Proportion of stroke patients anticoagulated during follow-up. | 3 months
  Proportion of patients prescribed with OAC as assessed at 3 month follow-up.
Rate of stroke recurrent, major adverse bleeding events and detection of AF outside the study protocol. | 1 year
  One year rate of recurrent ischemic stroke or TIA, hemorrhagic stroke, major adverse bleeding events and detection of AF outside the study protocol.
Time to first detection of AF or atrial flutter. | 7 days
  Time to first detection of AF or atrial flutter within 7 days of Holter monitoring.
Health Outcomes. | 1 year
  Health outcome as evaluated by Eq-5D Questionnaire.

OTHER OUTCOMES:
Predictors of occult AF. | 1 month
  To identify predictors of occult AF based on clinical, neuroimaging, echocardiography and Holter monitoring results.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hui Ping Foo, MD, Principal Investigator — Sarawak General Hospital
Locations (1):
- Sarawak General Hospital, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
The final decision is depending on the agreement among the co-investigators.